CLINICAL TRIAL: NCT03048838
Title: A Couple-based HIV Prevention Intervention to Promote HIV Protection Among Latino Male Couples
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Temple University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Columbia University (Other); Nova Southeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24120
Record Dates: First submitted 2017-02-03; First posted 2017-02-09 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to either risk-reduction group (Conectado Latinos en Parejas, CLP) or wellness-promotion (WP) control condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Risk reduction behavioral intervention (Experimental): Couples randomized to the risk reduction behavioral intervention ("Conectando Latinos en Pareja") will participate in four weekly sessions with a facilitator. Each session will last 2 hours. Participants will receive information and complete activities, participate in games and discussions to improve their relationship and improve health.
  Interventions: Behavioral: Risk reduction behavioral intervention
- Wellness Promotion Intervention (Active Comparator): Couples randomized to the wellness promotion control group will receive the same number of hours of attention as the active experimental group but will not receive the risk reduction intervention. Information presented will consist of topics related to general health.
  Interventions: Behavioral: Wellness Promotion Intervention

INTERVENTIONS:
Behavioral: Risk reduction behavioral intervention
  Arms: Risk reduction behavioral intervention
Behavioral: Wellness Promotion Intervention
  Arms: Wellness Promotion Intervention

SUMMARY:
Epidemiological studies have attributed the source of many new HIV and STI infections among MSM to primary partners. Despite recent emphasis on couples-based interventions, efficacious interventions for Latino male couples have yet to be tested. The proposed study builds on the PI's post-doctoral research in which he adapted evidence based intervention for Black MSM couples, Connect 'n Unite, for Latino male couples using methodologically rigorous adaptation procedures. The adapted intervention, Conectado Latinos en Parejas (CLP) expands the prevention alternatives offered in previous interventions by incorporating biomedical prevention methods such as pre-exposure prophylaxis (PrEP), promoting engagement in care, adherence to treatment regimens and viral suppression (TasP) and encouraging routine HIV testing if appropriate given the couple's serostatus. The investigators will conduct a randomized control trial (RCT) to examine whether participants assigned to CLP report an increase in the proportion of HIV protected anal sex acts (operationalized as using condoms, PrEP, TasP) compared to those assigned to a Wellness Promotion (WP) time matched attention control. The investigators will recruit 150 Latino male couples from the Philadelphia MSA and randomly assign them to CLP or WP. Participants will complete ACASIs to assess behavioral and psychosocial factors and be tested for sexually transmitted infections (STI) at baseline, 3 and 6 month post intervention. The investigators will conduct optional HIV/STI testing at baseline, 3, and 6 month post intervention. The primary study activities will be conducted at a large Latino serving CBO in North Philadelphia. To our knowledge, this study will be the first to examine the impact of a couple-based intervention to increase HIV protected anal sex acts for Latino male couples capable of being scaled up and replicated in various communities to provide continuous support and protection for this heavily impacted group.

DETAILED DESCRIPTION:
Latino men who have sex with men (MSM) continue to be disproportionately affected by HIV. Experiences of stigma, discrimination, marginalization, sexual objectification, negative cultural perceptions of homosexuality, and cultural values such as 'familismo' and 'machismo' elevate their vulnerability to HIV infection. Many Latino MSM use substances as a way to cope with or alleviate these stressors, further increasing their risk. Although efficacious interventions for Latino MSM have been developed, not a single one has focused on Latino male couples, despite strong evidence from White MSM that HIV infection often occurs within primary couple relationships. Findings from the investigators formative study with Latino MSM suggest that the factors driving HIV risk for White male couples also operate among Latino male couples. For instance, Latino men in male couples were more likely to report condomless anal sex and problematic alcohol use than those who were not in a relationship. Developing and testing tailored interventions for Latino male couples, as the investigators are proposing, is warranted.

The proposed study builds on the PI's post-doctoral research which adapted an evidence based intervention for Black MSM couples, Connect 'n Unite (CNU), for Latino male couples using methodologically rigorous adaptation procedures. The adapted intervention, Conectando Latinos en Pareja (CLP), expands the prevention alternatives offered in previous interventions by incorporating biomedical prevention methods such as pre-exposure prophylaxis (PrEP); promoting engagement in care, adherence to treatment regimens and viral suppression (TasP) for HIV-positive individuals and/or couples; and encouraging routine HIV testing, if appropriate given the couple's serostatus. The investigators have proposed a two-phase study to determine the preliminary efficacy of Conectando Latinos en Pareja to increase the proportion of anal sex acts that are HIV protected (i.e. anal sex acts in which condoms, PrEP, TasP, or combination thereof reduce risk of HIV transmission). During Phase 1, the investigators will develop and finalize the intervention manuals and assessment instruments, pilot test the intervention, and conduct the necessary preparatory activities for launching a randomized control trial (RCT). During Phase 2, the investigators will conduct a RCT to examine whether participants assigned to CLP report an increase in the proportion of HIV-protected anal sex acts compared to those assigned to a Wellness Promotion (WP), a time-matched attention control (the investigators will use an algorithm that incorporates use of condoms, PrEP, and/or TasP, depending on the serostatus of the couple to compute the dependent variable).

The investigators will recruit 150 Latino male couples (where at least one member of the dyad self-identifies as Latino) in the corridor between Philadelphia, PA and Trenton, NJ - an area with porous borders where many diverse subgroups of Latinos live. The investigators will randomly assign couples to CLP or WP. The investigators will assess sexual, alcohol and drug use behaviors and other psychosocial factors (e.g., depressive symptoms, anxiety symptoms) at baseline, 3, and 6 months post-intervention. Participants who consent to optional HIV/STI testing will be tested for HIV, chlamydia, and gonorrhea at baseline and at 3 and 6 months post-intervention. The primary assessment and project management activities will be conducted at GALAEI, a large Latino-serving CBO in North Philadelphia. Recruitment and screening will be done at community and internet venues. Intervention activities will be conduct at GALAEI, Temple University, and other safe spaces convenient to study participants.

ELIGIBILITY:
Inclusion Criteria:

1. be at least 18 years old;
2. report having a main/primary male partner during the past 90 days (operationalized as a man with whom he has had a sexual relationship during the past 90 days and has a strong emotional bond);
3. self-identify as Latino/Hispanic or identify as having a main partner who identifies as Latino/Hispanic;
4. reports sexual activity in the past 90 days as described in the screening instrument;
5. identify each other as their main partner;
6. able to speak English and/or Spanish;
7. plan to remain in the area for the next 8 months.

Exclusion Criteria:

Couples will be excluded if:

1. either partner reports that participating in a study that talks about sex, relationship issues and alcohol/drugs will put him in danger;
2. either partner has a language or cognitive impairment that would prevent comprehension of study procedures;
3. either partner is currently on PrEP and fully adherent, or enrolled in any other HIV prevention study;
4. either partner is planning to move outside the area in the next 8 months;
5. either partner is planning on ending the relationship with his partner in the next 8 months; and
6. either partner reports being in a stable triadic relationship (operationalized as a relationship in which all 3 men have a strong emotional bond and the 3 men are having sex with each other).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Enrollment will be limited to Latinos males and their same-sex partners
Enrollment: 300 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Change in proportion of HIV protected anal sex acts between baseline and six months | 6 months post-intervention
  Change in proportion of anal sex acts involving protective measures (condoms, PrEP, TasP) to reduce risk of HIV transmission between baseline and six months

CONTACTS AND LOCATIONS:
Overall Officials: Omar Martinez, JD, Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinez O, Isabel Fernandez M, Wu E, Carballo-Dieguez A, Prado G, Davey A, Levine E, Mattera B, Lopez N, Valentin O, Murray A, Sutton M. A couple-based HIV prevention intervention for Latino men who have sex with men: study protocol for a randomized controlled trial. Trials. 2018 Apr 5;19(1):218. doi: 10.1186/s13063-018-2582-y. PMID 29622045